CLINICAL TRIAL: NCT06359600
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HS-10501 Tablets After Single and Multiple Oral Doses in Healthy Subjects
Brief Title: A Study of HS-10501 Tablets in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-10501-101
Record Dates: First submitted 2024-03-21; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): Single dose of HS-10501 administered orally under fasted conditions
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 2 (Experimental): Single dose of HS-10501 administered orally under fasted conditions
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 3 (Experimental): Single dose of HS-10501 administered orally under fed and fasted conditions
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 4 (Experimental): Single dose of HS-10501 administered orally under fasted conditions
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 5 (Experimental): Single dose of HS-10501 administered orally under fasted conditions
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 6 (Experimental): Single dose of HS-10501 administered orally under fasted conditions
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 7 (Experimental): Drugs are given twice a day (BID) for 27 days, and only one morning dose is given on the 28th day.
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 8 (Experimental): Drugs are given once a day (QD) for 28 days.
  Interventions: Drug: HS-10501 tablet; Drug: Placebo
- Cohort 9 (Experimental): Drugs are given twice a day (BID) for 27 days, and only one morning dose is given on the 28th day.
  Interventions: Drug: HS-10501 tablet; Drug: Placebo

INTERVENTIONS:
Drug: HS-10501 tablet — Administered orally
Drug: Placebo — Administered orally

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, Pharmacokinetics and Pharmacodynamics of single dose and multiple dose of HS-10501 tables in healthy subjects. This is the first clinical study of HS-10501 tables. This study has 2 parts. Parts A involve a single dose of HS-10501 tables or placebo and will last about 8 days. Also, this part will also further explore the food effect. Parts B involve multiple doses of HS-10501 tables or placebo and will last about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol;
2. Must be 18 to 55 years of age (inclusive) healthy male or female;
3. Body weight of at least 50.0 kg for male, and 45.0 kg for female; and Body Mass Index (BMI) within the range of 19.0 to 28.0 kg/m2 (inclusive);
4. Subjects (including partners) of childbearing potential are willing to use protocol specified effective methods of contraception from the date of signing the informed consent form to 30 days after the last dose;
5. Female subjects must have a negative blood pregnancy test report 3 days before dosing.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Subjects with a history of cardiovascular, respiratory, liver, kidney, digestive tract, mental, neurological, hematological, immune, and metabolic abnormalities and other diseases, and not suitable for the study as assessed by the investigator;
3. Subjects with clinically significant abnormalities in vital signs, physical examination, laboratory tests, or 12-lead ECG during the screening period;
4. Have received major surgery within 3 months before screening or have surgery plan during the study;
5. History of severe infection within 30 days before screening or currently experiencing severe infection;
6. The alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) are higher than the upper limit of normal (ULN);
7. Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or treponema pallidum antibody (TP-Ab);
8. Glycosylated hemoglobin (HbA1c) ≥ 6.0% and fasting blood glucose ≤ 3.9 mmol/L (70 mg/dL) or ≥ 6.1 mmol/L (110 mg/dL) at screening;
9. History of drug abuse and use of hard drugs within 1 year before the study or positive for urine drug screening;
10. Addicted to smoking or smokers who smoke 5 or more cigarettes per day on average within 3 months before screening;
11. History of alcohol abuse, or a single consumption of more than 14 units of alcohol in the past two weeks, or positive for breath alcohol test at screening;
12. Participating in any clinical trial involving drugs or medical devices within 3 months before screening;
13. Blood donation or loss of ≥ 400 mL or blood transfusion within 3 months before screening; blood donation or loss of ≥ 200 mL within 1 month before screening;
14. Subjects with severe allergic disease, or suspected allergy to any ingredient in the study drugs, or allergic constitution;
15. Subjects with concomitant diseases that may significantly affect the absorption of drugs or nutrients as judged by the investigator;
16. Subjects with a history of pancreatitis, and serum amylase or lipase greater than the ULN;
17. History or family history of medullary thyroid cancer and multiple endocrine neoplasia syndrome type 2;
18. Diet or weight loss treatment within 3 months prior to administration or having weight change of more than 5% or significant change in living habits;
19. Any medication taken within 2 weeks or 5 half-lives (whichever is longer) before screening and any medication expected to be taken throughout the study;
20. Any physiological or psychological diseases or conditions that may increase the risk of the study, affect the subject's compliance with the protocol, or affect the subject's completion of the study, as judged by the investigator;
21. Those who should not be enrolled per the investigator's opinion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE) , serious AEs and AE leading to withdrawal from treatment. | Day1 to last follow-up, SAD: Baseline to Day 8; MAD: Baseline to Day 35.
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Number of participants with clinically significant abnormalities in lab tests | Day1 to last follow-up, SAD: Baseline to Day 8; MAD: Baseline to Day 35.
  Laboratory tests include blood routine, urine routine, blood biochemistry and coagulation function, etc.
Number of participants with clinically significant change from baseline in vital signs | Day1 to last follow-up, SAD: Baseline to Day 8; MAD: Baseline to Day 35.
Change from baseline in Electrocardiogram (ECG) | Day1 to last follow-up, SAD: Baseline to Day 8; MAD: Baseline to Day 35.
  ECG parameters including heart rate, PR interval, QRS interval and QTcF, etc.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of HS-10501 - AUC0-t | pre-dose to 72 hours post-dose
  Area under the concentration-time curve from time zero to the last quantifiable time point t (AUC0-t)
Pharmacokinetic (PK) profile of HS-10501 - AUC0-∞ | pre-dose to 72 hours post-dose
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞);
Pharmacokinetic (PK) profile of HS-10501 - Cmax | pre-dose to 72 hours post-dose
  Maximum observed concentration (Cmax)
Pharmacokinetic (PK) profile of HS-10501 - Tmax | pre-dose to 72 hours post-dose
  Time to maximum observed concentration (Tmax)
Pharmacokinetic (PK) profile of HS-10501 - t1/2 | pre-dose to 72 hours post-dose
  Terminal elimination half-life (t1/2)
Pharmacokinetic (PK) profile of HS-10501 - CL/F | pre-dose to 72 hours post-dose
  Apparent clearance (CL/F)
Pharmacokinetic (PK) profile of HS-10501- Vz/F | pre-dose to 72 hours post-dose
  Apparent volume of distribution (Vz/F)
Pharmacokinetic (PK) profile of HS-10501-λz | pre-dose to 72 hours post-dose
  elimination rate constant (λz)
Pharmacokinetic (PK) profile of HS-10501- AUC0-τ | pre-dose to 72 hours post-dose
  area under plasma concentration-time curve within a dosing interval
Pharmacodynamic (PD) profile of doses of HS-10501 - AUC0-t of blood glucose-time curve after oral glucose tolerance test (OGTT) | before to 3 hours after the first intake of glucose on Day-1，Day 1 and Day 28
  Area under the glucose-time curve from time zero to the last quantifiable time point t (AUC0-t) after oral glucose tolerance test (OGTT)
Pharmacodynamic (PD) profile of doses of HS-10501 - AUC0-t of blood insulin-time curve after oral glucose tolerance test (OGTT) | before to 3 hours after the first intake of glucose on Day-1，Day 1 and Day 28
  Area under the insulin-time curve from time zero to the last quantifiable time point t (AUC0-t) after oral glucose tolerance test (OGTT)
body weight changes | from day-1to day 28
  Change in body weight from baseline after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Anhui University, Hefei, Anhui, China